CLINICAL TRIAL: NCT06267482
Title: Challenging The TKA Standard Of Care: Patient Specific Surgical Targets As Enabled By The Rosa
Brief Title: Using ROSA for Challenging The TKA Standard of Care
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 122311
Record Dates: First submitted 2024-01-02; First posted 2024-02-20 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Standard of care medial parapetallar approach
- ROSA PSA Parapatellar Approach (Active Comparator): Arm using the ROSA with PSA and medial parapetallar approach
  Interventions: Procedure: ROSA PSA Parapatellar Approach
- ROSA PSA Subvastus Approach (Active Comparator): Arm using the ROSA with PSA and medial subvastus approach
  Interventions: Procedure: ROSA PSA Subvastus Approach

INTERVENTIONS:
Procedure: ROSA PSA Parapatellar Approach — This intervention will consist of using the ROSA alongside patient-specific alignment. The knee incision will be the same as the standard of care (medial parapatellar approach).
  Arms: ROSA PSA Parapatellar Approach
Procedure: ROSA PSA Subvastus Approach — This intervention will consist of using the ROSA alongside patient-specific alignment. The knee incision will be an alternative, quad-sparring, subvastus approach.
  Arms: ROSA PSA Subvastus Approach

SUMMARY:
This is a prospective, randomized controlled trial using the cruciate retaining, MC Persona to comparing the conventional TKA to ROSA assisted TKA. Patients will be randomized to one of three study trial arms.

1. Standard of care medial parapetallar approach (Control)
2. ROSA PSA medial parapetallar approach
3. ROSA PSA medial subvastus approach Participants will be followed for 1 year post surgery with a combination of perioperative parameters, imaging, patient reported outcomes, functional outcomes, blood and tissue sampling for inflammatory information and activity levels.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is performed to treat end-stage arthropathy of the knee with substantial increases in surgical volumes projected from the existing 750,000 surgeries performed in North America annually. The current standard of care for a primary TKA is a medial parapatellar exposure with the surgical objective of a mechanically neutral limb alignment, with the tibial component perpendicular to the anatomic axis of the tibia. As patient dissatisfaction in their TKA is substantial, surgeons, allied health care workers and patients continue to work to optimize the outcomes by tailoring surgical approaches to patient specific characteristics, with a goal to diminish early and post-operative causes of dissatisfaction. As patient-reported functional outcomes scores are an important contributor of dissatisfaction, understanding how surgical objectives and technology affect measurable functional outcomes, patient-reported outcomes, health economic and inflammatory response is important.

One of the developing thoughts in TKA surgery has been the elucidation of the range of native alignment of patients' anatomy. As placing TKA components in positions dictated by the patient's unique anatomy has garnered greater attention, literature has suggested that respecting the patient's native anatomy of joint alignment may result in equivalent or possibly improved functional outcome scores compared to neutral mechanical alignment. Simultaneously, concerns have been raised that substantial varus alignment will inadvertently occur, with resultant negative impact on longevity. A more directive patient specific alignment (PSA) concept is the anatomic alignment approach that is built around the objective of achieving a 3 degree varus joint line with respect to the mechanical axis of the leg. It is thought that this may improve patient satisfaction and function as the anatomy of the joint is preserved, including improved soft tissue balance with less soft tissue releases required. However, as conventional instrumentation is imprecise and its use can result in a range of component alignments, a surgical objective of slight varus has a substantial risk of having the implants in too great of joint line angulation resulting in reduced longevity. Improved surgical instrumentation is required to enable PSA with the objective of precisely attaining anatomic alignment to avoid the negative effect of overly varus alignment.

Zimmer-Biomet has introduced the unique ROSA orthopaedic robot. This surgical instrument will enable the surgeon to easily achieve surgical objectives with greater precision than conventional techniques. In contrast with the market leader in orthopaedic robotic assistance, the ROSA also enables the surgeon to be flexible with surgical approach and potentiate intraoperative decision making by providing greater information intra-operatively. It also enables image or imageless care pathways to enable surgeons to do surgical planning themselves to create unique surgical objectives for each patient. These market differentiating features of this orthopaedic robot advance orthopaedic care and provide the basis of expanding the orthopaedic community's understanding of PSA. The robot will also enable further challenges to the current standard of care TKA. For example, quadriceps sparing approaches such as the subvastus approach have been demonstrated to improve early functional recovery but has also been suggested to have higher rates of implant malalignment. The flexibility of approach as well as the precision of the ROSA will potentiate this approach for enhanced recovery programs, which are important in this time of increased health care burdens with limited resources as well as demands for outpatient procedures. Finally, as the Persona ® MC potentiates physiologic function of the knee with a medial pivot point rather than non-physiologic kinematics of many other TKA designs, the knee potentially will feel more physiologic. As objective and subjective functional outcomes are substantial contributors to patient dissatisfaction, understanding how patient specific alignment and soft tissue sparing approaches might improve functional outcome is critical. Wearable technology, another recent advancement within orthopaedics, has demonstrable ability to measure innumerable functional variables, and will enable a greater understanding of how the ROSA in combination with the Persona MC will lead to improved outcomes and reduced resource use.

Current literature has used inflammatory response to assess the decreased amount of soft tissue disruption after robotic versus conventional TKA. Since objective and subjective joint stiffness and reduced range of motion are common complaints among patients with suboptimal outcomes after TKA, The investigators will examine knee inflammation and fibrosis as these likely contribute to stiffness. Understanding the effect of PSA ROSA TKA with the Persona MC on local and systemic inflammation both early post-operatively as well as at one year post-operatively will be achieved by advanced imaging as well as systemic markers in the context of each individual patient's unique cellular characteristics. Our proposal will also enable quantification of how soft tissue preserving approaches affect the local inflammatory response as well as muscle atrophy or edema.

Patient reported outcome measures (PROMs) are an important subjective metric to measure surgical success and traditionally have been the primary outcome measure for many studies. However, PROMs are limited by the multi-factorial nature of the measure as well as limited responsiveness and substantial ceiling effect. The improved data collection of wearable technology has enabled differentiation of factors influencing patient satisfaction with smaller numbers of patients. Because of this, wearable technology has several advantages as a primary outcome, including the fact that wearable technology directly measures functional outcomes: a primary source of dissatisfaction after a TKA. As restoration of the patient's anatomy within defined limits should enable the implant to function with greater harmony within the envelope of static and dynamic soft tissues, functional outcomes will be the primary outcome of this proposed randomized control trial (RCT).

The investigators propose in this prospective RCT to randomize 90 patients to one of three trial arms. The control trial arm will be the standard of care TKA Persona MC and be compared to PSA ROSA TKA with the Persona MC experimental arms of two different surgical exposures. The purpose is to examine the trajectory of functional recovery as well as PROMs and inflammatory response of standard of care TKA compared to outcomes enabled by the ROSA with the objective of improving care for TKA patients.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis of the knee indicating primary total knee arthroplasty
* Varus knee deformity of 0 to 10 degrees
* Sufficient ligamentous function to warrant retention of the posterior cruciate ligament
* Between the ages of 21 and 80 inclusive
* Patients willing and able to comply with follow-up requirements and self-evaluations
* Ability to give informed consent

Exclusion Criteria:

* Active or prior infection
* Medical condition precluding major surgery
* Predominantly inflammatory arthropathy
* Patellectomy
* PCL deficiency
* Major coronal plane deformity
* Prior trauma to the tibia or femur resulting in malalignment, canal occlusion, or open reduction and internal fixation
* Valgus alignment
* Neurologic condition limiting mobility
* Bone defects requiring augments, cones and/or stemmed implants

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Functional Outcome - Weight-bearing CT scan | Pre-operation, 1-3 days post-op, 6-weeks post-op, and 1-year post-op
  Patients will undergo a weight-bearing CT scan to examine implant migration and bone position in the knee.
Functional Outcome - 3D Ultrasound | Pre-operation, 6-weeks post-op, 3-months post-op and 1-year post-op
  Patients will undergo a 3D Ultrasound to measure the inflammatory characteristics including Synovial fluid and synovial thickness for fibrosis in the supra-patellar region of the knee
Functional Outcome - Timed Up and Go test | Pre-operation, 6-weeks post-op, 3-months post-op and 1-year post-op
  Patients will undergo a Timed Up and Go (TUG) test. Patients will have to get up from a seated position, walk 10 feet, turn around and walk another 10 feet. This test is used to examine the function of the lower extremities. A time improvement of 2.27 Seconds will be considered clinically meaningful
Patient health status - Knee Society Score | Pre-operation, 6-weeks post-op, 3-months post-op and 1-year post-op
  This will be done by comparing the Knee Society Score (KSS) Patient-reported outcome measurement questionnaire given to patients. The KSS questionnaire looks at several factors such as patient satisfaction (scale from 1-5, 5 being the best), Patient expectation (scale from 1-5, 5 being the best) and patient's pain during activities (scale from No pain to severe pain)
Patient health status - EuroQuol Survey | Pre-operation, 6-weeks post-op, 3-months post-op and 1-year post-op
  This will be done by comparing the EuroQuol (EQ-5D) Patient-reported outcome measurement questionnaire given to patients. EQ-5D looks at the overall quality of life of a patient. The survey has 2 sections, the first asking the patient to best describe their health (Scale from Unable to perform the activity to no problem performing the activity) and an overall health assessment (scale 0-100, 100 being the best health you can imagine)
Patient health status - Knee Injury and Osteoarthritis Outcome Score | Pre-operation, 6-weeks post-op, 3-months post-op and 1-year post-op
  This will be done by comparing the Knee Injury and Osteoarthritis Outcome score (KOOS) Patient-reported outcome measurement questionnaire given to patients. The KOOS survey looks at the pain and function of the operated knee. Patients will be asked questions about the pain they feel during activities (Scale from none-extreme) and the function of their joint (scale from none-extreme)
Patient health status - Western Ontario and McMaster Universities Arthritis Index | Pre-operation, 6-weeks post-op, 3-months post-op and 1-year post-op
  This will be done by comparing the Western Ontario and McMaster Universities Arthritis Index (WOMAC) Patient-reported outcome measurement questionnaire given to patients. This survey will ask patients about the pain, stiffness and difficulty of using their knee. This survey is scaled from 0-4, 0 being none and 4 being extreme.
Patient health status - Global Assessment | Pre-operation, 6-weeks post-op, 3-months post-op and 1-year post-op
  This will be done by comparing the UCLA Activity Score (UCLA) Patient-reported outcome measurement questionnaire given to patients. This survey assesses the activity level of patients on a scale from 0 - 10 with 10 being the patient regularly participates in impact sports.

SECONDARY OUTCOMES:
Health Ecominics | Pre-operation, 1-3 days post-op, 6-weeks post-op, 3-months post-op
  Patients will be asked to fill out a cost-diary to determine if the new methods help reduce resource consumption

CONTACTS AND LOCATIONS:
Overall Officials: Brent Lanting, PhD, Principal Investigator — London Health Sciences Center
Locations (1):
- University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Abdel MP, Oussedik S, Parratte S, Lustig S, Haddad FS. Coronal alignment in total knee replacement: historical review, contemporary analysis, and future direction. Bone Joint J. 2014 Jul;96-B(7):857-62. doi: 10.1302/0301-620X.96B7.33946. PMID 24986936
- [Background] Lanting BA, Lieberman JR, Callaghan JJ, Berend ME, MacDonald SJ. Ensuring a Winner: The ABCs of Primary Total Knee Arthroplasty. Instr Course Lect. 2015;64:369-79. PMID 25745921
- [Background] Bourne RB, Chesworth BM, Davis AM, Mahomed NN, Charron KD. Patient satisfaction after total knee arthroplasty: who is satisfied and who is not? Clin Orthop Relat Res. 2010 Jan;468(1):57-63. doi: 10.1007/s11999-009-1119-9. PMID 19844772
- [Background] Dunbar MJ, Richardson G, Robertsson O. I can't get no satisfaction after my total knee replacement: rhymes and reasons. Bone Joint J. 2013 Nov;95-B(11 Suppl A):148-52. doi: 10.1302/0301-620X.95B11.32767. PMID 24187375
- [Background] Gunaratne R, Pratt DN, Banda J, Fick DP, Khan RJK, Robertson BW. Patient Dissatisfaction Following Total Knee Arthroplasty: A Systematic Review of the Literature. J Arthroplasty. 2017 Dec;32(12):3854-3860. doi: 10.1016/j.arth.2017.07.021. Epub 2017 Jul 21. PMID 28844632
- [Background] Noble PC, Conditt MA, Cook KF, Mathis KB. The John Insall Award: Patient expectations affect satisfaction with total knee arthroplasty. Clin Orthop Relat Res. 2006 Nov;452:35-43. doi: 10.1097/01.blo.0000238825.63648.1e. PMID 16967035
- [Background] Vandekerckhove PTK, Matlovich N, Teeter MG, MacDonald SJ, Howard JL, Lanting BA. The relationship between constitutional alignment and varus osteoarthritis of the knee. Knee Surg Sports Traumatol Arthrosc. 2017 Sep;25(9):2873-2879. doi: 10.1007/s00167-016-3994-4. Epub 2016 Feb 1. PMID 26831863
- [Background] Lanting BA, Williams HA, Matlovich NF, Vandekerckhove PJ, Teeter MG, Vasarhelyi EM, Howard JL, Somerville LE. The impact of residual varus alignment following total knee arthroplasty on patient outcome scores in a constitutional varus population. Knee. 2018 Dec;25(6):1278-1282. doi: 10.1016/j.knee.2018.08.019. Epub 2018 Oct 9. PMID 30314879
- [Background] Howell SM, Hodapp EE, Vernace JV, Hull ML, Meade TD. Are undesirable contact kinematics minimized after kinematically aligned total knee arthroplasty? An intersurgeon analysis of consecutive patients. Knee Surg Sports Traumatol Arthrosc. 2013 Oct;21(10):2281-7. doi: 10.1007/s00167-012-2220-2. Epub 2012 Oct 2. PMID 23052114
- [Background] Howell SM, Howell SJ, Kuznik KT, Cohen J, Hull ML. Does a kinematically aligned total knee arthroplasty restore function without failure regardless of alignment category? Clin Orthop Relat Res. 2013 Mar;471(3):1000-7. doi: 10.1007/s11999-012-2613-z. Epub 2012 Sep 21. PMID 22996362
- [Background] Howell SM, Papadopoulos S, Kuznik KT, Hull ML. Accurate alignment and high function after kinematically aligned TKA performed with generic instruments. Knee Surg Sports Traumatol Arthrosc. 2013 Oct;21(10):2271-80. doi: 10.1007/s00167-013-2621-x. Epub 2013 Aug 15. PMID 23948721
- [Background] Dossett HG, Estrada NA, Swartz GJ, LeFevre GW, Kwasman BG. A randomised controlled trial of kinematically and mechanically aligned total knee replacements: two-year clinical results. Bone Joint J. 2014 Jul;96-B(7):907-13. doi: 10.1302/0301-620X.96B7.32812. PMID 24986944
- [Background] Dossett HG, Swartz GJ, Estrada NA, LeFevre GW, Kwasman BG. Kinematically versus mechanically aligned total knee arthroplasty. Orthopedics. 2012 Feb 17;35(2):e160-9. doi: 10.3928/01477447-20120123-04. PMID 22310400
- [Background] Fang D, Ritter MA. Malalignment: forewarned is forearmed. Orthopedics. 2009 Sep;32(9):orthosupersite.com/view.asp?rID=42850. doi: 10.3928/01477447-20090728-29. PMID 19751003
- [Background] Moreland JR, Bassett LW, Hanker GJ. Radiographic analysis of the axial alignment of the lower extremity. J Bone Joint Surg Am. 1987 Jun;69(5):745-9. PMID 3597474
- [Background] Berend ME, Ritter MA, Meding JB, Faris PM, Keating EM, Redelman R, Faris GW, Davis KE. Tibial component failure mechanisms in total knee arthroplasty. Clin Orthop Relat Res. 2004 Nov;(428):26-34. doi: 10.1097/01.blo.0000148578.22729.0e. PMID 15534515
- [Background] Ritter MA, Davis KE, Meding JB, Pierson JL, Berend ME, Malinzak RA. The effect of alignment and BMI on failure of total knee replacement. J Bone Joint Surg Am. 2011 Sep 7;93(17):1588-96. doi: 10.2106/JBJS.J.00772. PMID 21915573
- [Background] Fang DM, Ritter MA, Davis KE. Coronal alignment in total knee arthroplasty: just how important is it? J Arthroplasty. 2009 Sep;24(6 Suppl):39-43. doi: 10.1016/j.arth.2009.04.034. Epub 2009 Jun 24. PMID 19553073
- [Background] Alcelik I, Sukeik M, Pollock R, Misra A, Naguib A, Haddad FS. Comparing the mid-vastus and medial parapatellar approaches in total knee arthroplasty: a meta-analysis of short term outcomes. Knee. 2012 Aug;19(4):229-36. doi: 10.1016/j.knee.2011.07.010. Epub 2011 Aug 20. PMID 21862334
- [Background] Liu HW, Gu WD, Xu NW, Sun JY. Surgical approaches in total knee arthroplasty: a meta-analysis comparing the midvastus and subvastus to the medial peripatellar approach. J Arthroplasty. 2014 Dec;29(12):2298-304. doi: 10.1016/j.arth.2013.10.023. Epub 2013 Oct 28. PMID 24295800
- [Background] Xu SZ, Lin XJ, Tong X, Wang XW. Minimally invasive midvastus versus standard parapatellar approach in total knee arthroplasty: a meta-analysis of randomized controlled trials. PLoS One. 2014 May 20;9(5):e95311. doi: 10.1371/journal.pone.0095311. eCollection 2014. PMID 24845859
- [Background] Thienpont E. Faster quadriceps recovery with the far medial subvastus approach in minimally invasive total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2013 Oct;21(10):2370-4. doi: 10.1007/s00167-012-2215-z. Epub 2012 Sep 25. PMID 23007414
- [Background] Schroer WC, Diesfeld PJ, Reedy ME, Lemarr AR. Surgical accuracy with the mini-subvastus total knee arthroplasty a computer tomography scan analysis of postoperative implant alignment. J Arthroplasty. 2008 Jun;23(4):543-9. doi: 10.1016/j.arth.2007.05.034. Epub 2007 Nov 7. PMID 18514872
- [Background] Kayani B, Tahmassebi J, Ayuob A, Konan S, Oussedik S, Haddad FS. A prospective randomized controlled trial comparing the systemic inflammatory response in conventional jig-based total knee arthroplasty versus robotic-arm assisted total knee arthroplasty. Bone Joint J. 2021 Jan;103-B(1):113-122. doi: 10.1302/0301-620X.103B1.BJJ-2020-0602.R2. PMID 33380182
- [Background] Vasarhelyi EM, Williams HA, Howard JL, Petis S, Barfett J, Lanting BA. The Effect of Total Hip Arthroplasty Surgical Technique on Postoperative Muscle Atrophy. Orthopedics. 2020 Nov 1;43(6):361-366. doi: 10.3928/01477447-20200910-01. Epub 2020 Sep 22. PMID 32956472
- [Background] Giesinger K, Hamilton DF, Jost B, Holzner B, Giesinger JM. Comparative responsiveness of outcome measures for total knee arthroplasty. Osteoarthritis Cartilage. 2014 Feb;22(2):184-9. doi: 10.1016/j.joca.2013.11.001. Epub 2013 Nov 18. PMID 24262431
- [Background] Bloomfield RA, Williams HA, Broberg JS, Lanting BA, McIsaac KA, Teeter MG. Machine Learning Groups Patients by Early Functional Improvement Likelihood Based on Wearable Sensor Instrumented Preoperative Timed-Up-and-Go Tests. J Arthroplasty. 2019 Oct;34(10):2267-2271. doi: 10.1016/j.arth.2019.05.061. Epub 2019 Jun 5. PMID 31255408